CLINICAL TRIAL: NCT07028346
Title: An Exploratory Study of the Relationship Between Substance Use, Sleep Disturbances and Reward Sensitivity - A Randomized Control Trial of Cognitive Behavioral Therapy for Insomnia
Brief Title: Exploring Substance Use, Sleep Disturbances and Reward Sensitivity
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kwai Chung Hospital (Other)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Fritz Yeung, Clinical Psychologist, Kwai Chung Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIRB-2025-173-4
Record Dates: First submitted 2025-06-11; First posted 2025-06-19 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Substance Abuse; Sleep Disturbances
Keywords: Substance abuse; substance misuse; sleep disturbances; sleep problem
MeSH Terms: conditions — Substance-Related Disorders; Parasomnias | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBTi Group (Experimental): Cognitive Behavioral Therapy for Insomnia
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Sleep Education Group (Active Comparator): Sleep Education
  Interventions: Behavioral: Sleep Education

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — Cognitive Behavioral Therapy for Insomnia (CBT-I) is a first-line, non-medication treatment for insomnia that helps individuals identify and change the thoughts and behaviors that contribute to their sleep problems.
  Arms: CBTi Group
Behavioral: Sleep Education — Sleep Education group comprises psychoeducation sessions on sleep hygiene.
  Arms: Sleep Education Group

SUMMARY:
According to foreign medical studies, substance use is closely related to reward sensitivity and sleep patterns. The purpose of this research is to understand the relationship between these three factors, which will help improve medical treatment and overall care for substance misuse in the future. Participants will be randomized into CBTi and sleep education groups, and their substance/ alcohol use, sleep parameters and reward sensitivity will be measured at multiple time points.

DETAILED DESCRIPTION:
The study will invite approximately 154 individuals who have misused alcohol or drugs in the past three months and have symptoms of insomnia to participate. After completing the screening, participants who meet the study criteria will be asked to fill out five additional research questionnaires and take a 15-minute computer-based reward sensitivity test. Participants will then be randomly assigned, in a 1:1 ratio, to one of the following groups:

1. A three-session cognitive behavioral therapy (CBT) group (the first session lasts 60 minutes, with subsequent sessions not exceeding 30 minutes) and two follow-up phone calls (each lasting around 20 minutes).
2. A three-session sleep education group (the first session lasts 60 minutes, with subsequent sessions not exceeding 30 minutes) and two follow-up phone calls (each lasting around 20 minutes).

All participants will be invited to complete additional research questionnaires and computer-based tests in the 4th and 8th weeks after the group sessions begin.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who receive treatment services at Substance Abuse Assessment Clinic and other psychiatric out-patient clinics of Kwai Chung Hospital;
2. Individuals who have problematic substance or alcohol use in the past 3 months, confirmed by scores higher than or equal to 1 in both part 1 and part 2 of Tobacco, Alcohol, Prescription medication, and other Substance use (TAPS);
3. Individuals who have sleep disturbances, confirmed by a score higher than or equal to 8 on the Insomnia Severity Index (ISI).

Exclusion Criteria:

1. Individuals who cannot understand Cantonese, or cannot read Traditional Chinese
2. Individuals who cannot provide informed consent due to, for example, intoxication or abnormal mental state
3. Individuals who report abnormal or unstable mental states, such as active psychotic symptoms or acute intoxication, at any point of the study
4. Individuals who work overnight or have rotating shifts
5. Individuals who report pregnancy or medical conditions (including sleep apnea) that may have a severe impact on sleep
6. Individuals who use hypnotics regularly

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-06-16 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Insomnia Severity Index | From enrollment to the end of treatment at 8 weeks
Pittsburgh Sleep Quality Index | From enrollment to the end of treatment at 8 weeks
Drug Use Disorders Identification Test | From enrollment to the end of treatment at 8 weeks
Alcohol Use Disorders Identification Test | From enrollment to the end of treatment at 8 weeks

SECONDARY OUTCOMES:
Sensitivity to Reward Scales from Sensitivity to Reward and Sensitivity to Punishment Questionnaire | From enrollment to the end of treatment at 8 weeks
  Scores ranges from 0 to 48. Higher scores indicate greater sensitivity to reward, suggesting an increased behavioral tendency toward reward-seeking stimuli.
Computerized Iowa Gambling Task | From enrollment to the end of treatment at 8 weeks

OTHER OUTCOMES:
Client Satisfaction Questionnaire (CSQ-8) | At the end of treatment at 8 weeks
  Scores ranges from 8 to 32. Higher scores reflect greater overall satisfaction with services received, indicating a more positive client experience.

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared because of organizational policy.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-05-29): https://cdn.clinicaltrials.gov/large-docs/46/NCT07028346/Prot_SAP_000.pdf